CLINICAL TRIAL: NCT04020991
Title: Sleepiness and Tiredness Among Doctors Working In A Tertiary Hospital: Is it Work Related or Is There Underlying Sleep Disorders
Brief Title: Sleepiness and Tiredness Among Doctors Working in A Tertiary Hospital
Status: Completed | Type: Observational
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Other Study IDs: 1
Record Dates: First submitted 2019-07-11; First posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Doctors working in a tertiary hospital: Doctors working in a tertiary hospital
  Interventions: Diagnostic Test: Sleep Study

INTERVENTIONS:
Diagnostic Test: Sleep Study — Participants who noted to have Oxygen Desaturation Index more than 10 (moderate to severe OSA) will be referred to do formal sleep study and referral to Sleep Medicine Clinic

SUMMARY:
Sleep disorders are important health issues that can reduced ones quality of life by affecting their performance and productivity in a negative way. People who work in shifts or doing 24 hours call usually have irregular sleep patterns and often complaint of fatigue and daytime sleepiness. This will jeopardized our attention, concentration ability and memory which may lead to serious job accidents. This study is to screen for obstructive sleep apnea among doctors working in a tertiary hospital and to determine the predictors of OSAS and tiredness among doctors who frequently work night shifts or 24 hour call.

What would this involve? Participant will be required fill up demographic data and answer the STOP-Bang and Epworth sleepiness scale questionnaires. After that participant will need to wear a wrist watch pulse oximeter just before going to sleep at night until the next morning (minimum of 6 hours of sleep required). The wrist watch will then be returned to researcher the following day for data analysis purpose.

The benefits We hope to screen and identify those who are at risk of having obstructive sleep apnea and start early treatment among doctor who often have irregular sleep patterns and insufficient sleep due to the nature and timing of their work.

DETAILED DESCRIPTION:
INTRODUCTION Sleep disorder is common health problem globally. There are still many adult with clinically significant sleep disordered breathing remained undiagnosed. The most common sleep disorder is obstructive sleep apnoea (OSA) which is a sleep related breathing disorder characterized by full or partial cessation in airflow that lasts more than 10 seconds despite a continuous effort to breath. It can occur due to recurrent collapsed or obstruction of the upper airway caused by relaxation of the uvula and soft palate which leads to a hallmark of snoring and gasping pattern. The blood oxygen levels will be reduced during this interruption of breathing that leads to occasional hypoxemia causing an individual to arouse from sleep a few times and hence ending with poor quality of sleep. The common symptoms experienced by individuals with OSA include fatigue, excessive daytime sleepiness (EDS), insomnia, nocturia and morning headaches.

Diagnosis of OSA is confirmed with a polysomnography (PSG). The total number of apnoea plus hypopnoea events divided by total sleep hours is the Apnoea-Hypopnoea Index (AHI). If the AHI is 5 times/ hour or greater, a diagnosis of OSA is made. Despite PSG being the gold standard in diagnosing OSA, due to resource limited settings, there are several screening questionnaires and clinical modalities that have been developed to assess the risk of having OSA. The snoring, tiredness, observed apnoea, high blood pressure, high BMI, age, neck circumference and male gender (STOP-Bang) questionnaire is an effective and concise screening tool which consist of eight dichotomous (Yes/No) questions. The total score range from 0-8. Patients with STOP-Bang score of 0 to 2 can be classified as low risk for moderate to severe OSA while midrange score 3-4 and score of 5-8 has intermediate and high risk for moderate to severe OSA respectively.

Epworth Sleepiness Scale (ESS) is the most commonly used questionnaire for measuring sleepiness via sleep propensity. The total ESS scores are based on eight different situational sleep propensities, which give an average sleep propensity. ESS values ranged from 0 (unlikely to fall asleep in any situation to 24 (high chance of falling asleep in all eight situations). ESS values of at least 10 were used to define excessive daytime sleepiness Nocturnal oximetry can be a simple alternative to polysomnography to detect sleep disordered breathing. Oxygen desaturation index (ODI) is the hourly average number of desaturations , which are defined at least 4% decrease in saturation from the average saturation in preceding 120 seconds, and lasting more than 10 seconds. Alternatively ODI is a good predictor of AHI. ODI >10 has a high sensitivity (93%) and reasonable specificity (75%) to detect moderate and severe sleep disorder breathing Sleep disorders are important health issues that can reduced ones quality of life by affecting their performance and productivity in a detrimental way. Trainee doctors who frequently work in night shifts or 24hours shift commonly have irregular sleep patterns and sleep deprivation causing sleepiness and tiredness. When insufficient sleep coexist with shift work, an increased tendency to sleep poses a more serious problem especially during work. This also causes deterioration in neurocognitive functions such as attention, concentration ability and memory which may lead to serious job accidents. The data on prevalence of sleep disorders among resident doctors are still limited. Hence, more research needed to evaluate if the sleepiness and tiredness among doctors were due to the nature of their work or is there underlying sleep disorders which may contribute to the symptoms of undiagnosed of OSA.

OBJECTIVE The primary objective of this study is to see the prevalence of OSA Syndrome among trainee doctors working in a tertiary hospital . Second objective is to identify predictors for OSAS, tiredness and perception of inadequate sleep in this study population.

MATERIALS AND METHOD This quantitative study with a prospective cross sectional method will be submitted for approval of research supervisor of Department of Anaesthesiology University Malaya Medical Centre (UMMC) and the Medical Research and Ethics Committee of University Malaya Medical Centre.

Written informed consent will be obtained from healthcare providers recruited into this study which will be conducted by researcher herself.

Inclusions criteria

1. Doctors working in a tertiary hospital Exclusions criteria

1. Individuals which already diagnosed with OSA and on treatment
2. Pregnancy

Methodology All doctors recruited will be required to fill up the demographic data, STOP-Bang and Epworth Sleepiness Scale questionnaires. A wristwatch pulse oximetry will be given to each participant for home nocturnal oxygen saturation monitoring during sleep. Participant will have to wear the wristwatch prior to sleep at night till the next day. The STOP-Bang and ESS scores will be compared and correlate with data collected from the wristwatch pulse oximetry.

STATISTICAL ANALYSIS

1. Sample Size Calculation To estimate prevalence of snoring and obstructive sleep apnoea among healthcare providers working in Department of Anesthesiology and Intensive Care Unit University Malaya Medical Centre we need 203 staff to achieve 3% precision in estimating prevalence which was 5% in previous study (Omur et al., 2014) (Using Sample size calculator for Prevalence Studies, Naing et al., 2006)
2. Statistical tests Demographic data will analysed using multiple linear regression. The prevalence of OSA syndrome among trainee doctors will compared using Chi-square test. A value of p<0.05 will be considered statistically significant. Logistic regression analysis will be used to identify the predictors for OSAS; tiredness and perception of inadequate sleep.

ELIGIBILITY:
Inclusion Criteria:

* Doctors working in a tertiary hospital

Exclusion Criteria:

* Pregnancy
* Already diagnosed with OSA

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All doctors working in a tertiary hospital
Sampling Method: Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of OSA among doctors working in a tertiary hospital | 10months
  To determine whether the sleepiness and tiredness among doctors is contributed by undiagnosed sleep disorders

SECONDARY OUTCOMES:
Predictors of tiredness, perception of inadequate sleep and OSA syndrome in doctors population | 10 months
  To look at prevalence of OSA among doctors

CONTACTS AND LOCATIONS:
Overall Officials: Chew Yin Wang, MBChB, Study Chair — University of Malaya
Locations (1):
- University Malaya, Petaling Jaya, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chung F, Abdullah HR, Liao P. STOP-Bang Questionnaire: A Practical Approach to Screen for Obstructive Sleep Apnea. Chest. 2016 Mar;149(3):631-8. doi: 10.1378/chest.15-0903. Epub 2016 Jan 12. PMID 26378880
- [Background] Yasin R, Muntham D, Chirakalwasan N. Uncovering the sleep disorders among young doctors. Sleep Breath. 2016 Dec;20(4):1137-1144. doi: 10.1007/s11325-016-1380-6. Epub 2016 Aug 17. PMID 27535070
- [Background] Arunsurat I, Luengyosluechakul S, Prateephoungrat K, Siripaupradist P, Khemtong S, Jamcharoensup K, Thanapatkaiporn N, Limpawattana P, Laohasiriwong S, Pinitsoontorn S, Boonjaraspinyo S, Sawanyawisuth K. Simplified Berlin Questionnaire for Screening of High Risk for Obstructive Sleep Apnea Among Thai Male Healthcare Workers. J UOEH. 2016 Sep;38(3):199-206. doi: 10.7888/juoeh.38.199. PMID 27627967
- [Background] Chung F, Liao P, Elsaid H, Islam S, Shapiro CM, Sun Y. Oxygen desaturation index from nocturnal oximetry: a sensitive and specific tool to detect sleep-disordered breathing in surgical patients. Anesth Analg. 2012 May;114(5):993-1000. doi: 10.1213/ANE.0b013e318248f4f5. Epub 2012 Feb 24. PMID 22366847
- [Background] Chung F, Subramanyam R, Liao P, Sasaki E, Shapiro C, Sun Y. High STOP-Bang score indicates a high probability of obstructive sleep apnoea. Br J Anaesth. 2012 May;108(5):768-75. doi: 10.1093/bja/aes022. Epub 2012 Mar 8. PMID 22401881
- [Background] Fahzwi A, Basheer H, Pateer M & Sharma S. 2017. Oxygen Desaturation Index For Diagnosing Obstructive Sleep Apnoea in Patients With Morbid Obesity. Thorax 72: A115